CLINICAL TRIAL: NCT05717621
Title: The DelVIN Trial - A Multicenter Phase I Trial Evaluating the Safety and Preliminary Efficacy of Local Decitabine Treatment of Human Papillomavirus (HPV)-Induced Vulvar Intraepithelial Neoplasia (VIN) Grade 2/3
Brief Title: Clinical Trial With Local Decitabine Treatment of HPV-Induced VIN Grade 2/3 (DelVIN)
Acronym: DelVIN
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViMREX GmbH (Industry)
Collaborators: Frankfurter Institut für Klinische Krebsforschung IKF GmbH am Krankenhaus Nordwest (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: V-001; 2022-001834-12 (EudraCT Number)
Record Dates: First submitted 2023-01-10; First posted 2023-02-08 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Vulvar Intraepithelial Neoplasia Grade 2; Vulvar Intraepithelial Neoplasia Grade 3
Keywords: vulvar intraepithelial neoplasia (VIN)

STUDY DESIGN:
Intervention Model Description: Clinical trial with a single arm (one-group), all eligible patients will receive treatment with VTD-101 ointment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Test Arm (Experimental): VTD-101 ointment
  Interventions: Drug: VTD-101 ointment

INTERVENTIONS:
Drug: VTD-101 ointment — Self-administration of VTD-101 ointment (Decitabine ointment)

SUMMARY:
This is a multicentre open labelled phase I trial evaluating the safety and preliminary efficacy of local decitabine treatment of human papillomavirus (HPV)-induced vulvar intraepithelial neoplasia (VIN) grade 2/3.

The main purpose and primary objective of the study is to determine the recommended phase 2 dose (RP2D) of VTD-101 ointment for the topical treatment of HPV-induced VIN grade 2/3. The RP2D is defined as the dose that is safe, tolerable and effective. Corresponding endpoints are the rate of patients experiencing at least one dose limiting toxicity (DLT) and the rate of patients with clinical complete or partial response (cCR/cPR) according to adapted RECIST criteria.

Secondary objectives are to further characterize the efficacy of topical treatment with VTD-101 ointment, to further evaluate the safety and tolerability of topical treatment with VTD-101 ointment, and to evaluate quality of life (QoL) in patients treated with VTD-101 ointment.

ELIGIBILITY:
Inclusion Criteria:

1. Having provided written informed consent
2. Women ≥ 18 years of age at the time of signing the written informed consent
3. Women with histologically confirmed vulvar intraepithelial neoplasia (VIN) grade 2 or 3 (also referred to as "high grade VIN" or "high-grade squamous intraepithelial lesions [HSIL]")
4. Uni- or multifocal VIN grade 2 or 3
5. Newly diagnosed or recurrent VIN grade 2 or 3
6. Women who refuse standard therapy, have not responded (or no longer respond) to standard therapy, have not tolerated standard therapy or for whom standard therapy is contraindicated
7. Evidence of HPV-induced etiology of the lesion(s) as indicated by the detection of p16INK4a overexpression as well as high-risk (HR) HPV DNA presence in the lesion(s)
8. Women of childbearing potential (WOCBP) must agree to use one highly effective contraceptive method during the treatment period and for at least 6 months after the last IMP administration
9. Ability of patient to understand the character and individual consequences of the clinical trial
10. In the investigator's judgement, is willing and able to comply with the study protocol

Exclusion Criteria:

1. Evidence for or suspicion of vulvar tumor invasion
2. History of vulvar cancer
3. Previous surgical (except biopsy) or medical procedures of the high-grade VIN within the past 4 weeks prior to treatment start
4. Neutropenia or thrombocytopenia
5. Known allergy or hypersensitivity against decitabine or any of the excipients contained in the formulation
6. Current or prior use of immunosuppressive medication within 14 days (3 months for azathioprine, methotrexate, and tofacitinib) before the first dose of VTD-101 ointment. The following are exceptions to this criterion:

   * Intranasal, inhaled or topical (outside the anogenital area) steroids
   * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
   * Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
7. Medical conditions associated with severe immunosuppression (e.g., acquired immune deficiency syndrome [AIDS])
8. Active infection within the anogenital tract (except for HPV)
9. Malignancies within 5 years prior to study inclusion with the exception of malignancies with a negligible risk of metastases or death (5-year OS > 90%) like ductal carcinoma in situ or basalioma
10. Evidence of any other disease, neurologic or metabolic dysfunction, physical examination finding or laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of the study medication, puts the patient at higher risk for treatment-related complications or may affect the interpretation of study results
11. Participation in another interventional clinical study ≤ 4 weeks prior to initiation of study treatment or participation in such a study at the same time as this study
12. Receipt of an investigational drug within 4 weeks prior to initiation of study treatment
13. Pregnancy or breast feeding or planning to become pregnant during the treatment period or during the 6 months following the end of treatment. Women of childbearing potential must have a negative serum pregnancy test result within 7 days prior to initiation of study treatment
14. Women of childbearing potential who are unwilling to agree to remain abstinent (refrain from heterosexual intercourse) or to use contraceptive methods that result in a failure rate of <1% per year during the treatment period and for at least 6 months after the last IMP administration

Other study protocol-defined in-/exclusion criteria could apply.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2023-03-28 (Actual); Primary Completion 2025-01-17 (Actual); Study Completion 2025-01-17 (Actual)

PRIMARY OUTCOMES:
Determination of the dose that is safe and tolerable (by the assessment of the rate of patients (%) experiencing at least one dose limiting toxicity (DLT)) as part of the determination of the recommended phase 2 dose (RP2D). | 28 days
  The primary safety endpoint defined as rate of patients experiencing at least one DLT, will be identified by observing frequency, relation to IMP treatment and severity of specific AEs.
Determination of the dose that is effective (by the assessment of the rate of patients (%) with clinical complete or partial response (cCR/cPR) according to adapted RECIST criteria) as part of the determination of the recommended phase 2 dose (RP2D). | 16 months
  The primary efficacy endpoint is defined as proportion (%) of patients who achieved clinical complete or partial response, as assessed by adapted RECIST criteria. (Clinical complete response (cCR) is defined as: Complete visual disappearance of the treated lesion(s) (i.e., 100% reduction in the sum of the longest diameter (SLD) among all treated lesions). Clinical partial response (cPR) is defined as: 30-99% reduction in the SLD among all treated lesions.

SECONDARY OUTCOMES:
Rate of patients (%) with pathological complete response (pCR) | 4 months
  The efficacy will be further characterized by the rate of patients experiencing a pathological complete response of the treated lesion(s) in percent (%).
Computer-based read-out of clinical response | 16 months
  The efficacy will be further characterized by a computer-based read-out of manually annotated total surface area of the lesions (mm2/cm2), which will be followed by grading according to adapted RECIST criteria (cCR: 100% reduction in lesion size, cPR: 30-99% reduction in lesion size, SD: 1-29% reduction in lesion size, PD: ≥20% increase in lesion size).
Molecular response | 4 months
  The efficacy will be further characterized by the molecular response defined as reduction of combined p16INK4a/Ki-67-positive cells within the lesion (or in the region of the initial location of the lesion in case of complete lesion disappearance) and defined as decrease of DNMT1 protein expression in HPV-transformed cells determined by immunohistochemistry.
Clearance of HPV infection in the reference lesion | 4 months
  The efficacy will be further characterized by the analysis of the clearance of HPV infection in the reference lesion, defined as the absence of HPV DNA of the HR-HPV type(s) detected at baseline.
Disease recurrence in patients | 16 months
  The efficacy will be further characterized by determining the presence of recurrent lesions in treated patients. Disease recurrence is defined as the reappearance of lesions that were previously subject to complete clinical response.
Onset of new lesions | 16 months
  The efficacy will be further characterized by determining the presence of new lesions in treated patients. Onset of new lesions is defined as the appearance of new lesion(s) at a distinct vulvar site (i.e., a site different from the treated site(s)).
Adherence to the treatment plan assessed by drug accountability and patient diaries | 4 months
  The efficacy will be further characterized by the adherence of patients to the treatment plan. This will be assessed by IMP drug accountability as well as by self-reporting by patients according to a standardized study-specific questionnaire (paper-based patient diary).
Further evaluation of safety and tolerability of the treatment by the assessment of adverse events (AEs) according to NCI CTCAE v5.0 | 16 months
  The safety and tolerability of the treatment will be further assessed with the help of frequency tables with the number and percentage of patients who experienced the AE by treatment and total. Additionally, AEs will be summarized by seriousness of AE, relationship to the IMP, and grading for all NCI CTC categories (CTCAE v5.0).
Evaluation of the quality of life (QoL) in patients treated with VTD-101 ointment with the help of the following corresponding endpoint: "VIN questionnaire" (QoL questionnaire modified and translated from [Lockhart et al. 2013]). | 4 months
  QoL as assessed by means of 29 questions within the "VIN questionnaire" will be summarized using descriptive statistics and changes before and after treatment at respective time points by treatment and total.

CONTACTS AND LOCATIONS:
Overall Officials: Elena-Sophie Prigge, Dr., Study Director — ViMREX GmbH
Locations (5):
- Germany (5):
  - Universitätsklinikum Augsburg, Klinik für Frauenheilkunde und Geburtshilfe, Augsburg, Bavaria
  - Medizinische Hochschule Hannover Klinik für Frauenheilkunde und Geburtshilfe, Hanover, Lower Saxony
  - St. Elisabeth Krankenhaus Köln, Klinik für Gynäkologie und Geburtshilfe, Cologne
  - Frauenarztpraxis Heussweg Hamburg, Hamburg
  - Dysplasiezentrum HH am Krankenhaus Jerusalem, Hamburg

IPD SHARING:
Plan to Share IPD: No